CLINICAL TRIAL: NCT00681629
Title: CARE II - Evaluation of Treatment Outcomes in Schizophrenic Patients Taking Part in the Integrated Care Program - a Single-country, Multi-centre Phase IV Study
Brief Title: Schizophrenic Patients in Integrated Care
Acronym: CARE II
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty finding eligible sites/patients; current situation in health policy cause negative effect on existing/planned contracts for integrated care program
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00048
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Integrated Care; Quetiapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine XR Alone (Experimental): Oral administration as 200 mg and 300 mg tablets allowing flexible dosing in 100 mg steps. Once daily in the evening. On day 1: 300 mg quetiapine XR, on day 2 : 600 mg, from day 3 onwards 400 to 800 mg at the centre-specific investigator´s discretion
  Interventions: Drug: Quetiapine XR
- Quetiapine XR With Integrated Care Program (ICP) (Experimental): Oral administration as 200 mg and 300 mg tablets allowing flexible dosing in 100 mg steps. Once daily in the evening. On day 1: 300 mg quetiapine XR, on day 2 : 600 mg, from day 3 onwards 400 to 800 mg at the centre-specific investigator´s discretion
  Interventions: Drug: Quetiapine XR; Other: Integrated Care Program (ICP)

INTERVENTIONS:
Drug: Quetiapine XR — 400-800 mg, oral, bid
  Other Names: Seroquel Prolong
Other: Integrated Care Program (ICP) — Integrated care program (ICP), this is a legally based integrated care program covered by a contract according to §§ 140 a-d SGB-V (SGB: social security code); The ICP is not exclusively designed for this phase IV trial. Participation in the ICP is possible anytime for each patient in whom the services are covered by the individual health insurance.
  Arms: Quetiapine XR With Integrated Care Program (ICP)

SUMMARY:
The purpose of the study is to investigate the well-being of schizophrenic patients treated with quetiapine XR combined with participation in the integrated care program compared to a treatment with quetiapine XR alone over a period of 18 month

ELIGIBILITY:
Inclusion Criteria:

* Patients with baseline SWN-K <=70
* Provision of signed informed consent
* Out-patients with schizophrenia, schizophreniform disorder or schizoaffective disorder, severe postpartum depressive disorders with psychotic symptoms and a minimum HAM-D cut off score of 20 points

Exclusion Criteria:

* Evidence of a clinical relevant disease, eg renal or hepatic impairment, significant coronary heart disease, hepatitis B or C, AIDS
* Patients with known cardiovascular disease or other condition predisposing to hypotension or family history of QT prolongation
* Patients who pose an imminent risk of suicide or danger to self or others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lambert, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf, Martinistr. 52, 20246 Hamburg, Germany
Locations (8):
- Germany (8):
  - Research Site, München, Bavaria
  - Research Site, Oranienburg, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Lüneburg, Lower Saxony
  - Research Site, Oldenburg, Lower Saxony
  - Research Site, Chemnitz, Saxony
  - Research Site, Berlin, State of Berlin
  - Research Site, Stolberg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period July 2008 to November 2008; Centre Dr. Lambert (Hamburg), Centre Dr. Dorn (Berlin)
Groups:
- Quetiapine XR With Integrated Care Program (ICP): Oral administration as 200 mg and 300 mg tablets allowing flexible dosing in 100 mg steps. Once daily in the evening. On day 1: 300 mg quetiapine XR, on day 2 : 600 mg, from day 3 onwards 400 to 800 mg at the centre-specific investigator´s discretion.
  Integrated Care Program (ICP) is a legally based integrated care program covered by a contract according to §§ 140 a-d SGB-V (SGB: social security code); The ICP is not exclusively designed for this phase IV trial. Participation in the ICP is possible anytime for each patient in whom the services are covered by the individual health insurance.
Period: Overall Study
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Started | 5 (It was planned to recruit 100 patient) | 2 (It was planned to recruit 100 patient)
Completed | 0 | 0
Not Completed | 5 | 2
Not completed — Study termination | 4 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Customized [Number; unit: Participants]
  18-65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Subjective Well-being in Patients Treated for Schizophrenia, Schizoaffective Disorder, Schizophreniform Disorder, Delusional Disorder or Psychotic Disorder Not Otherwise Specified Using the SWN-K (Subjective Well-being Under Neuroleptics) Scale
Description: The SWN-K is comprised of 20 questions, each of which is rated using a 6 point scale ranging from 1 (not at all) to 6 (very much). Possible scores range from 20-120, with higher scores implying higher subjective well-being.
Time Frame: 4 months
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Subjective Well-being Using the SWN-K (Subjective Well-being Under Neuroleptics Scale) Total Score
Description: as for outcome 1
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Symptomatic Outcome Using CGI-S (Clinical Global Impression-Schizophrenia) Scale
Description: With the CGI-S the rate of the severity of a patient's symptoms (positive, negative, cognitive, depressive and overall) using a scale ranging from 1 (normal, not ill) to 7 (among the most severely ill) is measured - higher scores implying higher severity.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Symptomatic Outcome Using the PANSS-8 Scales(Positive and Negative Symptoms) Scale Score
Description: The schizophrenic symptomatology will be measured by the Positive and Negative Syndrome Scale (PANSS) providing 8 items of which each is rated on a severity scale ranging from 1-7, (1= absent - 7 = extreme severe. higher scores implying higher severity.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: GAF (Global Assessment of Functioning) Scale Score
Description: The "GAF" is a numeric rating scale used by clinicians for assessment of the social, occupational, psychological functioning of adult patients. The scale represents a hypothetical continuum of mental health illness providing a descending scoring code from 100 until 0. Higher scores indicate better patient condition and performance.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: PSP (Personal and Social Performance) Scale Score
Description: The '(PSP" rating scale (100 until 0) used by clinicians for assessment of 4 main domains of functioning in adult patients acc. (a) socially useful activities including work and study, (b) personal and social relationships, (c) self-care, and (d) disturbing and aggressive behavior. Higher scores indicate better patient condition and performance.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: EQ-5D (European Quality of Life Questionnaire) Score
Description: The EQ-5D questionnaire is a generic measure of health status. It defines health in terms of five dimensions:1 (Mobility); 2 (Self-care); 3 (Usual activity); 4 (Pain/Discomfort); 5 (Anxiety/Depression).
  The minimum possible value is 5 (one point for each dimension) and the maximum possible values is 15 (3 points for each dimension). Each dimension has 3 levels of "severity"- "no problems, "some problems" and "extreme problems". Higher scores indicate more problems.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Vocational Occupational Index "VOC" Score
Description: The "VOC" index will assess the following 7 items: 1 fulltime gainful employment, 2 homemaker or student, 3 part-time gainful employment (20 hours per week or less), 4 retired, 5 full or part-time volunteer, 6 on medical or psychiatric leave of absence, 7 unemployed, whether or not expected to work. Results will be descriptively summarized. The VOC index will be completed at each visit. Difference from baseline of the index will be derived at each assessment
Time Frame: Up to 18 months (V1 Day 1, V2 Month 1, V3 Month 3, V4 Month 6, V5 Month 12, V6 Month 18)
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Assess Quality of Life Levels Using the Q-LES-Q-18 (Quality of Life Enjoyment and Satisfaction) Questionnaire
Description: Q-LES-Q-18 will allow to generate a general QoL-index which will be used for the analysis and is defined as the average of the single scores for all 18 items. Scoring will be carried out from 1-5 per item (never / rarely / sometimes / frequently / all the time). Results will be descriptively summarized.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Assess Quality of Life Levels Using the RSM Scale (Riedel-Spellmann-Musil) Scale
Description: The '(RSM" is a new 36-item measure validated to assess the "QoL" in different dimensions of schizophrenic patient treated with antipsychotics. It will be rated on a four-point Likert scale (not / rather not / rather yes / yes) by the patient and the investigator. The total score ranges from min. 0 to max. of 108. Higher scores indicate higher "QoL".
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Assess Patient Engagement to Therapy Using the SES Scale (Service Engagement Scale)
Description: The 'SES" is a 14-item measure consisting of statements that assess the client specific engagement with services. It will be rated on a four-point Likert scale (not at all / rarely / sometimes / most of the time) by the investigator. The total score ranges from min. 0 to a max. of 42. Higher scores indicate lower engagement.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Assess Compliance/Medication Adherence Using the MARS Scale (Medication Adherence Rating Scale)
Description: The 'Medication Adherence Rating Scale' (MARS) is a reliable and valid self-reporting tool for investigation of the compliance in psychiatric patients also recognizing the complexity of compliance behaviour. 10 questions on medication attitude have to be answered by 'yes' or 'no' (8 times 1= no and Yes = 0 and twice 1= no, Yes =1). Results will be descriptively summarized. Summarized results minimum 0: low medication adherence, maximum 10: high medication adherence.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Number; unit: Participants
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Evaluate the Level of the Patients' (Subjective) Satisfaction Using the CSQ-8 Scale (Client Satisfaction Questionnaire)
Description: The 'CSQ-8" is a brief, self-administered method to monitor the consumer's satisfaction with services in outpatient psychotherapy, showing high internal consistency. It is identified as a core subset of the general CSQ covering 8 Likert-type items with four response choices where '1' indicates the lowest and '4' the highest degree of satisfaction.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Assess Health Economy Improvements in Terms of a Reduction in Treatment Costs and Loss of Productivity by Determination of the Total Cost by Number of Days With Hospitalization
Description: Any hospitalisation days in inpatients units and emergency ward stays will be recorded. At each hospitalisation, the number of days will be computed and at each visit, the cumulative total number of days will be used to calculate total costs. As higher the number of hospitalisation days as higher the costs per patient.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Assess Health Economy Improvements in Terms of a Reduction in Treatment Costs and Loss of Productivity by Determination of the Total Number of Days the Patient Was Not Able to Work or go to School or Complete Routine Daily Activities
Description: The number of lost work days, lost school days or days without completing routine daily activities will be evaluated. With any number of lost workdays or lost school days or without completing routine daily activities, the costs will increase and the productivity will decrease.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Assess Health Economy Improvements in Terms of a Reduction in Treatment Costs and Loss of Productivity by Determination of the Need for Any Additional Antipsychotic Medication
Description: Concomitant psychotropic drugs will be coded (ATC = Drug code) to allow a comparison of the number of drugs used per ATC class and per treatment visit. The drugs used will be listed by keeping their brand name for allowing to translate them into costs.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: Drugs
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Evaluate Safety and Tolerability by Evaluation of Weight/Waist Circumference
Description: Measuring of weight and waist circumference in centimeter.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Evaluate Safety and Tolerability by Evaluation of Laboratory Tests
Description: Measuring of: B-Haemoglobin (g/dl), B-Haematocrit(%), B-Erythrocyte count(pl), B-Leucocytes count (nl), B-Platelet count(nl), Complete blood count (nl), B-Leucocytes differential count (%), B-HbA1c(%), S-ALAT (U/l), S-ASAT (U/l), S-GGT (U/l), P-Glucose (fasting)(mh/dl), S-prolactin level (ng/ml), S-Pregnancy test (IU/l), Qualitative analysis of urine with Stix®,Urine pregnancy. Comparing results with standard values.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Mean (Full Range); unit: depending on the Lab test (see above)
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Evaluate Safety and Tolerability by Evaluation of Concomitant Medication
Description: Listing of all concomitant medication to show the efficacy and safety.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Number; unit: Name of concomitant medication
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Evaluate Safety and Tolerability by Evaluation of the Incidence of Adverse Events
Description: Listing of all adverse event or SAE´s to show the safety and tolerability.
Time Frame: 4 month
Population: No data were reported as no participants completed the study
Measure: Number; unit: number of events
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Quetiapine XR With Integrated Care Program (ICP) | Quetiapine XR Alone
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 2/5 | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Quetiapine XR With Integrated Care Program (ICP) (N=5) | Quetiapine XR Alone (N=2)
Fatigue (General disorders) | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Weight Increased (Investigations) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Abnormal Dreams (Psychiatric disorders) | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The study was stopped due to poor enrollment and no data analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site has to inform sponsor about a publication at least 60 day in advance and 10 days before submission of an abstract or presentation. Change requests by the sponsor are recognized unless the scientific character or the objectivity is on risk. If the sponsor plans a patent application the publication has to be postponed up to 120 days.